CLINICAL TRIAL: NCT02536391
Title: A Phase 1, Single-Dose, Randomized, Cross-Over, Relative Bioavailability, and Food Effect Study of Ipatasertib (GDC-0068) in Healthy Subjects
Brief Title: Ipatasertib (GDC-0068) Study to Evaluate Formulation Change and Food Effect on Bioavailability in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GO29868
Record Dates: First submitted 2015-08-27; First posted 2015-08-31 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — ipatasertib; Capsules; Tablets

ARMS (6):
- Sequence 1: Tablet/Capsule/Tablet with food (Experimental): Day 1: ipatasertib tablet administered after fast, Day 8: ipatasertib capsule administered after fast, Day 15: ipatasertib tablet administered after high-fat meal.
  Interventions: Drug: Ipatasertib (capsule); Drug: Ipatasertib (tablet)
- Sequence 2: Tablet/Tablet with food/Capsule (Experimental): Day 1: ipatasertib tablet administered after fast, Day 8: ipatasertib tablet administered after high-fat meal, Day 15: ipatasertib capsule administered after fast.
  Interventions: Drug: Ipatasertib (capsule); Drug: Ipatasertib (tablet)
- Sequence 3: Capsule/Tablet/Tablet with food (Experimental): Day 1: ipatasertib capsule administered after fast, Day 8: ipatasertib tablet administered after fast, Day 15: ipatasertib tablet administered after high-fat meal.
  Interventions: Drug: Ipatasertib (capsule); Drug: Ipatasertib (tablet)
- Sequence 4: Capsule/Tablet with food/Tablet (Experimental): Day 1: ipatasertib capsule administered after fast, Day 8: ipatasertib tablet administered after high-fat meal, Day 15: ipatasertib tablet administered after fast.
  Interventions: Drug: Ipatasertib (capsule); Drug: Ipatasertib (tablet)
- Sequence 5: Tablet with food/Tablet/Capsule (Experimental): Day 1: ipatasertib tablet administered after high-fat meal, Day 8: ipatasertib tablet administered after fast, Day 15: ipatasertib capsule administered after fast.
  Interventions: Drug: Ipatasertib (capsule); Drug: Ipatasertib (tablet)
- Sequence 6: Tablet with food/Capsule/Tablet (Experimental): Day 1: ipatasertib tablet administered after high-fat meal, Day 8: ipatasertib capsule administered after fast, Day 15: ipatasertib tablet administered after fast.
  Interventions: Drug: Ipatasertib (capsule); Drug: Ipatasertib (tablet)

INTERVENTIONS:
Drug: Ipatasertib (capsule) — Orally administered single dose of Ipatasertib formulated as a capsule.
  Other Names: GDC-0068 (capsule)
Drug: Ipatasertib (tablet) — Orally administered single dose of Ipatasertib formulated as a tablet.
  Other Names: GDC-0068 (tablet)

SUMMARY:
This Phase I, open-label, randomized, 3-period crossover study was designed to determine the relative bioavailability of ipatasertib administered as capsule and tablet formulations to healthy volunteers. In addition, the influence of food on ipatasertib exposure will also be determined. Participants will be randomized to one of six treatment sequences to receive three treatments of a single oral administration of ipatasertib in, 1) tablet formulation in the fasted state, 2) capsule formulation in the fasted state or 3) tablet formulation in the fed state. Pharmacokinetics will be assessed, and standard physical and clinical evaluations will be performed throughout the study. Time on study is expected to be 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females, between 18 and 55 years of age, inclusive
* Body mass index between 18.5 and 29.9 kg/m^2, inclusive

Exclusion Criteria:

- Clinically significant findings from medical history or screening evaluations.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of Ipatasertib | Days 1, 8 and 15
Time to Maximum Concentration (tmax) of Ipatasertib | Days 1, 8 and 15
Area Under the Concentration-time Curve (AUC) from Hour 0 to the Last Quantifiable Concentration (AUC0-t) of Ipatasertib | Days 1, 8 and 15
Area Under the Concentration-time Curve (AUC) from Hour 0 Extrapolated to Infinity | Days 1, 8 and 15
Apparent Terminal Elimination Half-Life (t1/2) of Ipatasertib | Days 1, 8 and 15
Apparent Total Clearance (CL/F) of Ipatasertib | Days 1, 8 and 15
Apparent Volume of Distribution (Vz/F) of Ipatasertib | Days 1, 8 and 15

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events | From check in (Day -1) to 30 days after the last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Madison, Wisconsin, United States

REFERENCES:
- [Derived] Malhi V, Budha N, Sane R, Huang J, Liederer B, Meng R, Patel P, Deng Y, Cervantes A, Tabernero J, Musib L. Single- and multiple-dose pharmacokinetics, potential for CYP3A inhibition, and food effect in patients with cancer and healthy subjects receiving ipatasertib. Cancer Chemother Pharmacol. 2021 Dec;88(6):921-930. doi: 10.1007/s00280-021-04344-9. Epub 2021 Sep 1. PMID 34471960